CLINICAL TRIAL: NCT00734461
Title: A Single-Center, Randomized, Double-Blind, Active- and Placebo-Controlled Crossover Study to Evaluate the Subjective Effects of PTI-801 in Non-Physically Dependent Subjects With a History of Drug Abuse
Brief Title: Study to Evaluate the Subjective Effects of PTI-801 in Non-Physically Dependent Subjects With a History of Drug Abuse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pain Therapeutics (Industry)
Responsible Party: Sponsor
Organization: PainT (Unknown)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PTI-801-XM
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-03

CONDITIONS: Opioid-Related Disorders
Keywords: Non-physically dependent subjects; history of opioid abuse
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Oxycodone; Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- Placebo (Placebo Comparator): Placebo, single dose
  Interventions: Drug: oxycodone and naltrexone
- Oxycodone 20 mg (Active Comparator): Oxycodone 20 mg single dose tablet
  Interventions: Drug: oxycodone and naltrexone
- Oxycodone 40 mg (Active Comparator): Oxycodone 40 mg single dose tablet
  Interventions: Drug: oxycodone and naltrexone
- PTI-801 20/.001 mg (Experimental): Oxycodone 20 mg / Naltrexone 0.001 mg
  Interventions: Drug: oxycodone and naltrexone
- PTI-801 40/.001 mg (Experimental): Oxycodone 40 mg / Naltrexone 0.001 mg
  Interventions: Drug: oxycodone and naltrexone
- PTI-801 20/.0001 mg (Experimental): Oxycodone 40 mg / Naltrexone 0.0001 mg
  Interventions: Drug: oxycodone and naltrexone
- PTI-801 40/.0001 mg (Experimental): Oxycodone 40 mg / Naltrexone 0.0001 mg
  Interventions: Drug: oxycodone and naltrexone

INTERVENTIONS:
Drug: oxycodone and naltrexone — tablets containing 20 mg or 40 mg oxycodone
  / tablets containing 20 mg or 40 mg oxycodone combined w/0.001 mg or 0.0001 mg naltrexone

SUMMARY:
This is a single-center, randomized, 7-way crossover, double-blind, active and placebo-controlled study to evaluate the subjective effects of oxycodone combined with ultra-low dose naltrexone in comparison to oxycodone alone in non-physically dependent subjects with a history of opioid abuse. Approximately 14 subjects will be randomized to one of fourteen sequences selected from a balanced 7x7 Latin square design and its mirror image.

DETAILED DESCRIPTION:
At the conclusion of a screening period, qualifying subjects with a negative urine drug screen and ethanol breath test will be admitted to an inpatient research unit. After a 24 hour observation period confirming that the subject is not undergoing opioid withdrawal, subjects will randomly receive either 30 mg oxycodone or matching placebo over two consecutive days in a double-blind fashion. The purpose of this oxycodone vs. placebo qualifying period is to select for subjects with a positive drug liking response and to orient subjects to the various scales. Only subjects with a positive response on the visual analog "Liking" scale of at least 20 points higher on active oxycodone vs. placebo will be eligible to continue in the double-blind 7-way crossover study. Fourteen subjects will be randomized to one of fourteen sequences.

Each subject will receive a single dose of one of the following 7 treatments:

Placebo, oxycodone 20 mg, oxycodone 40 mg, oxycodone 20 mg/naltrexone 0.001 mg, oxycodone 40 mg/naltrexone 0.001 mg,oxycodone 20 mg/naltrexone 0.0001 mg, oxycodone 40 mg/naltrexone 0.0001 mg.

Oxycodone and naltrexone will be formulated in combination as a single tablet. All tablets will be identical in appearance. The identity of each treatment will be unknown to all study personnel and subjects.

Immediately prior to and at specified time points after administration of a single dose of study drug, subjects will complete the following subjective scales: visual analog scales (VAS) for any drug effect, high, good effects, bad effects, liking, and sick; and adjective ratings (agonist and antagonist scales). Subjects will also be asked to complete a money versus drug questionnaire at various time points after drug administration. Observers will complete an adjective rating scale. Safety will be monitored by vital signs (heart rate, blood pressure, respiratory rate, and pulse oximetry), adverse events assessments, clinical laboratory tests, physical examinations and electrocardiograms (ECGs). In addition, pupil diameter (measured by photographs) will be obtained to monitor for physiological signs of opioid effects.

The first double-blind dose of study drug will be administered at least 24 hours after the last dose of the two day qualifying period. Dosings will be separated by a washout period of at least 120 hours (see sample calendar in Section 6.5). The observation period for safety will continue for 24 hours following the final dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Males and females who are at least 18 and no more than 65 years of age.
* The subject is in good health as determined by medical history and physical examination.
* The subject is willing and able to speak, read, and understand English and provide written informed consent.
* The subject's urine drug screen and ethanol breath test are negative at check-in to the clinic.
* The subject has a history of polydrug abuse and: Has taken illicit opioids within the last 30 days; and/or Misused/abused prescription opioids within the last 30 days.
* The subject is willing and able to comply with all testing and requirements defined in the protocol.
* The subject must agree to refrain from caffeine and xanthine-containing products throughout the study, and to refrain from nicotine from 1 hour prior to each dosing until 4 hours after each dosing.
* The subject is willing and able to remain at the study site unit for the duration of the study.
* The subject has a positive response to oxycodone in the blinded qualifying period as defined by a VAS Liking score for oxycodone that is at least 20 points greater than that for placebo.
* Females who are postmenopausal, physically incapable of childbearing, or practicing an acceptable method of birth control. Acceptable methods of birth control include surgical sterilization, hormonal contraceptives, or double-barrier methods (condom or diaphragm with a spermicidal agent or intrauterine device [IUD]). A negative pregnancy test result must be obtained for all females at screening and at check-in to the clinic.

Exclusion Criteria:

* The subject has a positive urine drug screen or ethanol breath test at check-in to the clinic.
* The subject has been taking prescription opioids daily for chronic pain or has been taking illicit or prescription opioids daily for recreational purposes for more than 20 days in the last month.
* The subject is enrolled in treatment for drug abuse or is actively seeking treatment for drug abuse.
* The subject has any significant deviations from normal in physical examination, electrocardiogram (ECG), or clinical laboratory tests, as evaluated by the investigator.
* The subject has had a clinically significant illness within 30 days preceding entry into this study.
* The subject has a history of significant neurological, hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, or metabolic disease.
* The subject has a history of an allergic reaction to oxycodone or structurally similar compounds (morphine, hydromorphone, hydrocodone, levorphanol, pentazocine, codeine, etc.), naltrexone or other narcotic agonists.
* The subject has used any prescription medication (besides hormonal contraceptives) or recreational drugs within 7 days or over-the-counter (OTC) medication within 48 hours of check-in to the clinic or intends to use any prescription, recreational drugs or OTC medication during the study that may interfere with the evaluation of study medication.
* The subject has used alcohol, grapefruit, or grapefruit juice 24 hours before check-in to the clinic or intends to use any of these products during the study.
* The subject is pregnant or breastfeeding.
* The subject has received an investigational drug within 30 days prior to initiation of this study.
* The subject exhibits signs/symptoms of opioid withdrawal during the 24-hour observation period after check-in.
* The subject has a history of hospitalization due to a psychiatric disorder within the previous year or a current major psychiatric disorder. (Substance abuse disorders are not exclusionary).
* The subject experiences any of the following within 4 hours after administration of oxycodone 30 mg during the blinded qualifying dosing period: adverse events requiring narcotic antagonist administration, emesis, or opioid toxicity (see Section 10.0).
* The subject is unwilling to reside in the study unit for the inpatient portion of the study or to cooperate fully with the investigator or site personnel.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-08; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to evaluate the subjective effects of PTI-801 formulated with either 0.001 mg naltrexone or 0.0001 mg naltrexone compared to oxycodone alone in individuals with a history of opioid abuse. | At 30, 60, 90, 120, 150, 180 and 210 minutes post-dose

SECONDARY OUTCOMES:
Secondary objectives include determining the safety and physiological effects of single doses of PTI-801 compared to oxycodone following oral administration in individuals with a history of opioid abuse. | At 30, 60, 90, 120, 150, 180 and 210 minutes post-dose

CONTACTS AND LOCATIONS:
Overall Officials: George E Bigelow, PhD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States